CLINICAL TRIAL: NCT02735616
Title: Comparing the Behavior of the Cardiac Autonomic Regulation System During 24h in Patient Post Stroke and Controls
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, AVITAL HERSHKOVITZ, Avital Hershkovitz, Rabin Medical Center
Other Study IDs: 008215rmc
Record Dates: First submitted 2016-03-07; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Stroke
Keywords: heart rate variability; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- study: 15 CVA patients, 1-3 weeks after their first stroke. The patients will be hospitalized in the neurology department at the geriatric "Beit-Rivka" hospital at Petah-Tiva, Israel.
  patients with pacemaker or those who use Beta-Blocker drugs, as well as patients with cerebellar injury, will be excluded from the research
- control: 15 patients from the orthopedic department at the same hospital, matching by age and gender to the study group.

SUMMARY:
By Investigating the heart rate variability (HRV) of 15 patients after stroke and compare it to the HRV of 15 orthopedic patients, the investigators hope to achieve 3 main goals:

1. To describe the 24-hour circadian rhythm of heart rate among patients after stroke in the sub-acute phase during 3 days. 2. To examine the differences in the circadian rhythm of heart rate along 3 days between patients after stroke in the sub-acute phase and control group matched by age and gender. 3. To describe the reaction and examine the differences in reactions of the heart autonomic system during rest, paced breathing and activity in both groups- stoke and control.

The HRV will be monitored by Polar watch and the activity will be measured by accelerometer, both will be attached to the patients at the beginning of the trial and will stay on them for 3 whole days.

DETAILED DESCRIPTION:
Background: Evaluating the autonomic system is conducting, among others, by comparing the relationships between the two sub-systems that assembler it: the sympathetic and the parasympathetic systems. In normal conditions, there is balance between both systems which reflects in a highly dynamic heart rate and heart rate variability. As part of the brain injury after stroke, the autonomic system is also damaged. The heart rate variability is decreased and the 24-hour circadian rhythm of heart rate changes.

Purposes of the research: 1. To describe the 24-hour circadian rhythm of heart rate among patients after stroke in the sub-acute phase during 3 days. 2. To examine the differences in the circadian rhythm of heart rate along 3 days between patients after stroke in the sub-acute phase and control group matched by age and gender. 3. To describe the reaction and examine the differences in reactions of the heart autonomic system during rest, paced breathing and activity in both groups- stoke and control.

Methods:

Population: 15 patients after cerebrovascular accident (CVA), 1-3 weeks after the stroke. The patients will be hospitalized in the neurology department at the geriatric "Beit-Rivka" hospital. The control group will be 15 patients from the orthopedic department of the hospital' matching by age and gender. Tools: monitoring heart rate and heart rate variability by Polar watch (Polar RS800CX heart rate monitor). Monitoring activity will measure by accelerometer. Methods: after attaching to RS800CX watch, each participant will complete two tests: the response of heart rate to deep breathing and the response of heart rate variability to prolonged hand grip. The department nurse will be asked to answer a questionnaire regarding autonomic functions and the examiner will asses the functional independence of the participant by the "Functional Independence Measure" (FIM). In the research group will be additional assessments regarding the motor function by the "Stroke Activity Scale" and the "Scandinavian Stroke Scale". The watch and the accelerometer will stay on the participant for 3 day (72 hours) and the records regarding the daily activity such as meals, sleep, and all kind of treatments will be taken from the department's diary. At the end of three days, the data will be collected and analyzed on computer software.

ELIGIBILITY:
Inclusion Criteria:

* First stroke
* 1-3 weeks after the stroke

Exclusion Criteria:

* Pacemaker
* Cardiac arrhythmia
* Use of Beta- Blocker drugs
* Cerebellar deficit
* Mini-Mental State Examination (MMSE) < 18

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 CVA patients that are hospitalized in the neurology department at the geriatric "Beit-Rivka" hospital in Israel.
  The control group will be 15 patients from the orthopedic department of the hospital, matching by age and gender
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
heart rate variability | 3 days
  Heart rate variability will be measured by Polar watch at the beginning of each day during the 3 days of the research. At the end of those days, the data will be collected and analyzed on computer software.
step counter | three days follow up, (24-hours X 3)
  Step counter by Polar loop. Stored in the device and transfer to a computer for analysis.

SECONDARY OUTCOMES:
Stroke activity Scale | At admission
  A 5 items scale who measures the motor function at the level of disability in stroke patients. The functions included are getting out of bed, static and dynamic sitting balance, sitting to standing, stepping and walking and bringing a glass to the mouth.
Scandinavian Stroke Scale | At admission
  A 9 items scale (consciousness; eye movements; arm motor power; hand motor power; leg motor power; orientation; speech; facial palsy and gait) to assess neurological status.
Functional Independence Measure | At admission
  18 items scale designed to assess the amount of assistance required for a person with a disability to perform basic life activities safely and effectively. The activities include a mini- mum set of skills related to self-care, sphincter control, trans- fers, locomotion, communication, and social cognition.
Autonomic function questionnaire | At admission
  Based on the Svedberg questionnaire, originally made for children with cerebral palsy (CP) to describe symptoms such as cold extremities, constipation, pain, sleeping disorders and impaired well-being

IPD SHARING:
Plan to Share IPD: No